CLINICAL TRIAL: NCT00479778
Title: An Open Label, Randomized, Multicenter Study To Compare Bazedoxifene Steady-State Exposures Obtained With 2 Bazedoxifene Acetate/Conjugated Estrogen Formulations In Postmenopausal Women
Brief Title: Study Of Pharmacokinetic (PK) Profile of Bazedoxifene (BZA) in 2 BZA/Conjugated Estrogen Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3115A1-1121
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Postmenopause
Keywords: Postmenopause
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Bazedoxifene/conjugated estrogens

SUMMARY:
The purpose of the study is to understand how bazedoxifene is absorbed in the body when it is given in combination with 2 different formulations of conjugated estrogens. It is an open label study with no placebo control or comparator drugs. Subjects will take one dose of the investigation formulation daily for 14 days.

ELIGIBILITY:
* Postmenopausal women, aged 40 to 65 years.
* Use of oral estrogen-, progestin-, or androgen-, or SERM-containing drug products within 8 weeks before screening.
* A history or active presence of clinically relevant important medical disease.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72
Dates: Start 2007-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Gainesville, Florida, United States